CLINICAL TRIAL: NCT03004807
Title: Role of Centrum® Silver® in Improving Micronutrient Status in Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Tory Hagen, Professor, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: WI211838; 7158 (Other: Oregon State University IRB)
Record Dates: First submitted 2016-12-08; First posted 2016-12-29 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Vitamin Deficiency; Mineral Deficiency; Aging
Keywords: Nutrition; Aging; Multivitamin
MeSH Terms: conditions — Avitaminosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multivitamin (Experimental): Centrum Silver Men's Formula Multivitamin/Multimineral Supplement: 1/day
  Interventions: Dietary Supplement: Centrum Silver Mens' Formula
- Control (Placebo Comparator): Matching tablet to active multivitamin arm: 1/day
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Centrum Silver Mens' Formula — Multivitamin/Multimineral dietary supplement produced for Pfizer for use in older men.
  Other Names: Centrum Silver Men
  Arms: Multivitamin
Other: Control — A matching tablet to the dietary supplement, but without any active ingredients
  Other Names: Placebo Comparator
  Arms: Control

SUMMARY:
Older adults are susceptible to vitamin and mineral deficiencies for a variety of reasons and have an increased demand for many of these micronutrients. Multivitamin/multimineral supplement offer a simple way for adults to improve nutrient intake, but their ability to measurably affect micronutrient status in older adults has never been explored. This study intends to recruit healthy, non-smoking men aged 65 years or older. After meeting entry criteria, subjects will be required to restrict the use of supplements and/or fortified foods. Two months after these restrictions have begun, subjects will come to the clinical research center to take cognitive tests, undergo activity monitoring, provide blood samples for nutrition testing, and take food frequency questionnaires. Subjects will then be randomized into one of two groups - one consuming a multivitamin/multimineral supplement (Centrum Silver Mens Formula); another consuming an inert placebo tablet. Subjects will consume 1 tablet each day for six months. After this period, subjects will return to the clinical research center and repeat cognitive tests, activity monitor, blood sampling, and food frequency questionnaires. These data will be assessed to determine if multivitamin consumption results in changes in various nutrients versus taking a placebo (primary outcomes), and may results in changes lipid and lipoprotein profiles, metabolic health, inflammation, blood pressure or cognitive function (secondary outcomes). The investigators expect that results of this study will add to the general understanding if multivitamin/multimineral formulas can improve nutrition status of older adults, and therefore have the capacity of altering markers of health.

DETAILED DESCRIPTION:
Older adults are at increased risk of various chronic diseases, in which inadequate levels of vitamins and minerals may play a significant role, including cardiovascular disease, Alzheimer's disease, liver disease, and cancer. Most adults in the United States do not meet the Recommended Dietary Allowance (RDA) or Adequate Intake (AI) of many vitamins and nutritionally-essential minerals from diet alone, including vitamins A, C, D, E and K, calcium, magnesium, and potassium. Older adults are particularly susceptible to micronutrient inadequacies because of limited absorption, increased requirements, or - in the case of vitamin D - decreased synthetic capacity in the skin. Thus, there is a strong rationale for supplementing the diets of older adults with a multivitamin/multimineral supplement, such as Centrum® Silver®. However, little is currently known about the bioavailability of the Centrum® Silver® formula in this age demographic.

Epidemiological studies and recent clinical trials have shown that use of multivitamin/mineral supplements has beneficial effects on disease risk in men, including those of advanced age. It is assumed that these benefits of multivitamin/mineral supplements are achieved through changes in nutrition status. However, it has never been documented if there are concomitant changes in micronutrient levels in individuals who consume these supplements. Furthermore, changes in nutritional status in older individuals taking multivitamin/multimineral supplements are a subject that has yet to be explored.

Therefore, this study seeks to recruit men who are in generally good health, 65 years of age or older, to assess their vitamin and mineral status before and after six months (approximately 24 weeks) of supplementation with Centrum® Silver®. The investigators hypothesize that consuming multivitamin/multimineral supplements everyday will result in measurable increases in the status of one or more vitamins or minerals in the body. Concentrations of several vitamins and minerals in blood samples will be performed, along with a general assessment of micronutrient status in white blood cells (primary outcomes). To see if these changes in nutrition status impact other aspects of human health, changes in lipid and lipoprotein profiles, antioxidant status, metabolic health, and inflammation and treatment differences in cognitive function will be assessed (secondary outcomes). Centrum® Silver® supplementation may or may not have any effect on these secondary outcomes, when compared to a placebo, unless there are measurable changes in the primary outcomes.

The expectation is that the results of this research will add to a general understanding of multivitamin/mineral supplements and how well they can improve the nutritional status of older adults. By employing direct and functional methods to assay for nutritional content, this study will determine how well these methods correlate and by using both assay methods unique insight into the mechanism(s) whereby multivitamin/multimineral supplements might or might not lead to improvements in health may be ascertained.

ELIGIBILITY:
Inclusion Criteria:

Participants must be willing to:

* Consume a multivitamin/mineral supplement or placebo tablet each day during the 6-month study period
* Fill out online food frequency questionnaires
* Refrain from taking vitamin and mineral supplements that match micronutrients found in Centrum Silver (including certain antacids, energy drinks, fortified cereals, or nutritional shakes) other than those provided during the study. . Current users of supplements must agree to stop taking these supplements for two months before the study begins.
* Wear an activity monitor about the wrist continuously for two one-week periods, except when exposed to water, before and during multivitamin supplementation.
* Give blood samples on 3 separate occasions
* Participate in cognitive testing procedures

Exclusion Criteria:

* Currently taking supplements as recommended/ordered by a physician to correct a nutritional deficiency, with an exception for vitamins or minerals not found in Centrum Silver (as outlined in a Post-Screen Drug and Supplement Review).
* Current or recent (two years) history of smoking (tobacco or marijuana)
* Dysphagia or difficulty swallowing.
* Bariatric (gastric bypass) surgery or serious chronic illness that might affect absorption of multivitamins or minerals such as Crohn's disease, unmanaged celiac disease, chronic diarrhea, ulcerative colitis, gastritis, or a diagnosis of malabsorption syndrome.
* A diagnosis of cancer with chemotherapy or radiation treatment during the previous 5 years.
* Major surgery in the past 6 months or planned major surgery during the duration of the study.
* Prior heart attack, stroke, or heart failure.
* Uncontrolled stage II hypertension (blood pressure above 159/99 mm Hg).
* A current diagnosis of kidney, liver, or thyroid disease.
* Diabetes (Type 1 or Type 2).
* History of hypoglycemia or low blood sugar.
* Hb1ac levels > 6.4%.
* Fail a Post-Screen Drug and Supplement Review.
* BMI < 18.5 or > 35
* History of psychological or neurological disorders, or a diagnosis of dementia.
* Head injury with loss of consciousness of > 5 minutes in the last 5 years.
* Chronic Migraines - More than fifteen headache days per month over a three-month period of which more than eight are migraines.
* Score < 26 on the mini-mental state exam.
* Present treatment for drug or alcohol problems.
* Habit of taking three or more alcoholic drinks per day.
* Corrected visual acuity worse than 20/50.
* Anyone who cannot handwrite a letter or move a computer joystick with one of their hands.
* Cannot hear well enough to understand spoken instructions.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Plasma and Blood Cell Vitamin and Mineral Levels | Between baseline (visit 3) and 6 months after intervention begins (visit 7)
  Blood samples will be collected at baseline and end of intervention. Plasma levels of beta carotene, pyridoxine (vitamin B6), cobalamin (vitamin B12), ascorbic acid (vitamin C), 25-hydroxy vitamin D, α- tocopherol (vitamin E), and phylloquinone/menaquinones (vitamin K) will be determined. Analyses will be performed for absolute values and values corrected for total lipids where necessary. Folate will be assessed in red blood cells. Minerals analysis by inductively coupled plasma atomic emission spectroscopy (ICP-AES) will be performed in plasma or lymphocytes.

SECONDARY OUTCOMES:
Lipid Status | Between baseline (visit 3) and 6 months after intervention begins (visit 7)
  Changes to fasting lipoprotein and triglyceride status
High Resolution Respirometry | Between baseline (visit 3) and 6 months after intervention begins (visit 7)
  Isolated white blood cells will be evaluated in the Oroboros Oxygraph (Innsbruck, Austria) to evaluate the capacity of mitochondria to sustain respiration/energy demands
Cognitive abilities | Between cognitive baseline (visit 2) and 6 months after intervention begins (visit 6)
  Cognitive abilities will be assessed by the following NIH Toolbox measures: Picture Vocabulary, Flanker Inhibitory Control and Attention Test, Sorting Working Memory Test, Dimensional Change Card Sort Test, Pattern Completion Processing Speed Test, Picture Sequence Memory Test, and Oral Reading Recognition Test. The individual test scores are based on time and accuracy, will be normalized to scaled scores, and averaged to obtain a Fluid Cognition Composite score, as calculated by the NIH Toolbox scoring algorithms. Significant changes in total score after intervention, or between intervention and control groups will be recorded. Logical Memory will be tested with recall of narrative story both immediate and delayed as described in Wechsler Memory Scale-IV Protocol. Additionally, a "Head-Toes-Knees-Shoulders Task" that combines physical activity with processing speed and accuracy will also be assessed at the completion of each session.
Spatial memory as assessed by a virtual water maze | At visit 6, approximately 6 months after intervention begins, 1 week before visit 7
  A computerized environment will be presented for the subject that can be navigated with a joystick. The goal is to find a hidden platform based on spatial clues. Search accuracy for the target platform in the environment will be assessed between trials. Changes in proximity to the platform will be compared between successive trials in an individual, and also between individuals in the placebo control and multivitamin intervention groups.
Crystallized cognitive abilities | 1 week before intervention begins (visit 2) and 1 week before intervention ends (visit 6)
  Crystallized abilities will be assessed with NIH Toolbox Oral Reading Recognition Test and NIH Toolbox Picture Vocabulary Test. The individual test scores will be determined after adjusting for computer adaptive testing, normalized to scaled scores, and averaged to obtain a Crystallized Cognition Composite score, as calculated by the NIH Toolbox scoring algorithms. Significant changes in total score after intervention, or between intervention and control groups will be recorded.

OTHER OUTCOMES:
Activity Monitoring | Between visit 2 and visit 3 (duration: 1 week) and visit 6 and visit 7 (duration: 1 week)
  Wrist activity monitors (FitBit, commercial model) will be worn by subjects at the given intervals. General activity level, calories burned, heart rate, and steps taken will be recorded to give a general assessment of "energy level".

CONTACTS AND LOCATIONS:
Overall Officials: Tory M Hagen, PhD, Principal Investigator — Oregon State University
Locations (1):
- Linus Pauling Science Center, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in study data may contact the study principal investigators to request access. Data requests must be submitted in writing for approval by qualified individuals and will be reviewed by study investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study completion
Access Criteria: Project proposal form sent to the Linus Pauling Institute

REFERENCES:
- [Background] Michels AJ, Butler JA, Uesugi SL, Lee K, Frei BB, Bobe G, Magnusson KR, Hagen TM. Multivitamin/Multimineral Supplementation Prevents or Reverses Decline in Vitamin Biomarkers and Cellular Energy Metabolism in Healthy Older Men: A Randomized, Double-Blind, Placebo-Controlled Study. Nutrients. 2023 Jun 9;15(12):2691. doi: 10.3390/nu15122691. PMID 37375594